CLINICAL TRIAL: NCT04136301
Title: The Effect of Exposure to an Informative Video Regarding Possible Obstetric Emergencies on Maternal Anxiety and Peripartum Satisfaction- A Randomized Controlled Trial
Brief Title: The Effect of Exposure to an Informative Video on Maternal Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0093-19-WOMC
Record Dates: First submitted 2019-09-01; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Anxiety; Labor Pain; Patient Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Labor Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informative video arm (Experimental): Nuliparus women admitted to an induction will be exposed to informative video with data regarding labor and possible obstetric emergencies such as cesarean delivery.
  All patients will answer the State-Trait Anxiety Inventory (STAI) before and after intervention
  Interventions: Other: Informative Video group
- control arm (No Intervention): no intervention. All patients will answer the State-Trait Anxiety Inventory (STAI) before and after delivery.

INTERVENTIONS:
Other: Informative Video group — Informative Video group before labor in nulliparous women
  Arms: Informative video arm

SUMMARY:
Stress and anxiety during childbirth have negative consequence on both mother and fetus. Previous studies have learned the effect of several intervention to reduce anxiety during labor- such as music and foot reflexology. Nevertheless, data for informative video before labor for reducing stress and anxiety are sparse. The present study aimed to review and determine the effect of informative video on anxiety, pain and outcomes of the labor in primigravida women.

DETAILED DESCRIPTION:
A randomized control trial studying the effect of exposure to an informative video regarding labor and possible obstetrics emergencies on maternal anxiety and postpartum satisfaction

ELIGIBILITY:
Inclusion Criteria:

above 18 years of age Nulliparus women Informed consent Reads and understand Hebrew >37 weeks of gestation

Exclusion Criteria:

Refuse to participate Contraindications for vaginal delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 152 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory score in delivery room | 1 hour
  STAI questionnaire before and after delivery room

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No